CLINICAL TRIAL: NCT04490304
Title: How Durable is the Posterior Soft Tissue Repair After Total Hip Arthroplasty in Primary Osteoarthiritis Patients?
Brief Title: The Analysis of Posterior Soft Tissue Repair Durability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/252
Record Dates: First submitted 2020-07-25; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Arthroplasty Complications
Keywords: posterior soft tissue repair

STUDY DESIGN:
Intervention Model Description: prospective randomised trial
Masking Description: the x-ray measurements after the surgery were done by a care provider, not by the investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- posterior soft tissue repair durability (Other)
  Interventions: Other: durability of posterior soft tissue repair

INTERVENTIONS:
Other: durability of posterior soft tissue repair — how durable is the posterior soft tissue repair after total hip arthroplasty in primary osteoarthiritis patients?

SUMMARY:
Dislocation after THA usually occurs early after surgery and some go on to disabling recurrent dislocations . The posterior surgical approach is frequently used since it provides excellent exposure of both acetabulum and femur. However, many series on primary THA have reported that dislocation is 2 to 3 times more frequent after the posterior approach as compared to other approaches . Dissatisfaction with these dislocation rates resulted in the introduction of different posterior soft tissue repair techniques. Many authors have reported statistically significant differences in dislocation rates with posterior soft tissue repair as compared to without . However, there is still a concern in the literature regarding the durability of posterior soft tissue repair.

The aim of our study was to analyse THA patients with posterior soft tissue repair in terms of suture durability of two different suture materials and time of suture failure.

DETAILED DESCRIPTION:
A total of 42 consecutive THA patients (20 women,22 men) operated for primary osteoarthritis (OA) between 2018 and 2019 were included in the study. All patients were operated by the same orthopaedic surgeon under spinal anaesthesia via posterior approach using the same type of uncemented Polar stem(Smith and Nephew Inc) with 36 mm head in combination with uncemented Ep-Fit acetabular cup (Smith and Nephew Inc). All the patients were randomly divided into two groups. The randomization process was done by the odd and even number technique in which the patients with even inpatient numbers were assigned in Group A while the odd inpatient number patients were allotted in Group B. Patients in whom number 5 Ethibond Excel(Ethicon, Somerville, NJ) were used for soft tissue repair were included in Group A (n=22), whereas patients treated with number 2 Vicryl (Ethicon, Somerville,NJ)were in Group B (n=20).

The short external rotators tendons were released from the greater trochanter just at their insertion point. The capsule was incised, but not excised. The posterior repair included reattaching the piriformis,conjoined tendons and the capsule to the greater trochanter at the insertion point through 2, 2 mm drill holes with 2 stitches with non-absorbable no.5 Ethibond suture in one group and with absorbable no 2 vicryl suture in the other group after the prosthesis had been implanted and the joint reduced. One hemoclip was attached to the piriformis tendon and another to the conjoined tendons before pulling the sutures out of the drill holes in the trochanter. The suture materials lateral to the drill holes at the trochanter were also attached with two hemoclips.(fig 1-2) The postoperative regimen included walking with full weight bearing the next day after the surgery with a walking frame and without limitations in internal rotation or flexion. Anteroposterior radiographic examination was undertaken immediately after the patients returned from the operating theatre to the intensive care unit,at the 15th day, at 3 months and 6 months postoperatively (figure 3). The detachment of the hemoclips were measured during the follow up period.

ELIGIBILITY:
Inclusion Criteria:

primary osteoarthritis patients between 40-80 years old undergoing total hip replacement surgery between 2018-2019

Exclusion Criteria:

Any type of secondary osteoarthritis patients, and patients younger than 40 and older than 80 years old.

Ages: 41 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
elongation of capsular repair | 6 months
  measurement of detachment of the sutures after capsular repair

CONTACTS AND LOCATIONS:
Overall Officials: erdem edipoglu, Principal Investigator — Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Locations (1):
- Bakırkoysadikonuk, Istanbul, Bakırkoy, Turkey (Türkiye)